CLINICAL TRIAL: NCT04522440
Title: Natural Virtual Reality in the Application of Hospice Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 108110-F
Record Dates: First submitted 2020-08-11; First posted 2020-08-21 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Natural Virtual Reality in the Application of Hospice Care
Keywords: Natural virtual reality; hospice care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inpatients in hospice Ward (Experimental): Inpatients in hospice Ward with pain control problems
  Interventions: Other: to relieve the pain of inpatients in the hospice Ward

INTERVENTIONS:
Other: to relieve the pain of inpatients in the hospice Ward — This study will use pain scale, distress thermometer and POMS to understand whether the patient's pain status have changed.

SUMMARY:
In recent years, the use of Virtual Reality devices or somatosensory technology in various fields of teaching or sports has gradually matured. It is even possible to see that libraries or museums use virtual reality to promote reading or art. The trend of cross-border application has been born. The use of horticultural therapy in the current service of dementia or hospice patients is more common than in the past. The research team of the Taiwan Normal University has developed the first 3D Virtual Reality horticultural therapy course in Taiwan. Therefore, this study attempts to use natural virtual reality as an auxiliary care method to see if it can relieve the pain of hospitalized patients in the hospice ward, or relieve the stress of the caregiver (such as the patient's family or ward medical staff)!

The purpose of the study is:

1. Use natural virtual reality as an auxiliary care mode to relieve the painful condition of inpatients in the hospice ward.
2. Use natural virtual reality to relieve the psychological pressure of caregivers (family, medical colleagues).

The subjects of the study were: inpatients in the hospice ward of the hospital, caregivers of inpatients in the hospice ward, and medical staff of the hospice team.

Research methods:

1. Use virtual reality head-mounted equipment to watch the natural landscape for 10 minutes each time. The patient and caregiver watched three times a week during hospitalization. The medical staff watched eight times a day on weekdays.
2. Questionnaire: The patient used the pain scale and the Distress Thermometer (DT) scale as the pre-test questionnaire. The caregiver and the medical staff use the DT scale and the "Profile of Mood States (POMS)" as the pre-test questionnaire.

Expected results: The patient is expected to reduce the pain and enhance the quality of life by viewing the virtual natural landscape. It is expected that caregivers and medical colleagues can relieve stress and enhance the quality of life by watching virtual natural landscapes.

ELIGIBILITY:
Inclusion Criteria:

*Target: Inpatients in hospice Ward, carers of inpatients in hospice Ward, nurses or physicians of hospice team.

Exclusion Criteria:

* Due to the use of virtual reality headsets, people with eye diseases (glaucoma or cataracts and other people who are sensitive to light) and people with a history of mental illness are excluded.
* Inpatients in the hospice Ward also excluded those with tumors or diseases above the neck, those with symptoms of delirium, confusion, and unconsciousness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain scale | up to 2 weeks
  A single question, divided into 0-10 pain assessment scale.

SECONDARY OUTCOMES:
Distress Thermometer, DT | up to 2 weeks
  A single question, the height of emotional stress ranges from 0-10.

OTHER OUTCOMES:
POMS | up to 2 weeks
  The scale is divided into seven factors: vitality, self-esteem, confusion, fatigue, anger, tension and tension, with 37 items in total.

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Yi Lin, Principal Investigator — Family Medicine Department
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Banciao Dist, Taiwan

IPD SHARING:
Plan to Share IPD: No